CLINICAL TRIAL: NCT06505525
Title: Combined Intra- and Extra-articular ACL Reconstruction Versus Isolated Intra-articular ACL Reconstruction: Prospective Multicenter Randomized Clinical Trial With Hamstring Autograft
Brief Title: Combined Intra- and Extra-articular ACL Reconstruction Versus Isolated Intra-articular ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marcos Vinicius Credidio, Federal University of São Paulo, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1297-1650
Record Dates: First submitted 2024-06-03; First posted 2024-07-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Rupture; Ligament Knee Injury
Keywords: Rupture; Anterior Cruciate Ligament; Anterior Cruciate Ligament Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rupture

STUDY DESIGN:
Intervention Model Description: Prospective Multicenter Randomized Clinical Trial
Masking Description: Blinding after the assignment of patients to their group will be done as follows:
  * Participants: No blinding.
  * Investigators: No blinding.
  * Intervention providers: No blinding.
  * Data recorders: Partial blinding.
  * Outcome assessors: No blinding.
  * Data analysts, statisticians: Blinding. The statistician will only know the group of each patient after the statistical analysis is complete.
  * Care providers: No blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anatomical ACL reconstruction combined with extra-articular reconstruction with ALL (Experimental): Anatomical ACL reconstruction combined with extra-articular reinforcement reconstruction with ALL
  Interventions: Procedure: Extra-articular reconstruction with the Anterolateral Ligament
- Isolated intra-articular anatomical ACL reconstruction (Active Comparator): Isolated intra-articular anatomical ACL reconstruction
  Interventions: Procedure: Extra-articular reconstruction with the Anterolateral Ligament

INTERVENTIONS:
Procedure: Extra-articular reconstruction with the Anterolateral Ligament — Anatomical ACL reconstruction combined with extra-articular reconstruction with the Anterolateral Ligament

SUMMARY:
Abstract

Introduction: Autologous hamstring tendons are the most commonly used grafts in ACL reconstruction worldwide. There are several ways to prepare the graft using these tendons. One can prioritize increasing the diameter of an isolated intra-articular graft or alternatively, using one graft limb as an extra-articular reinforcement via the anterolateral ligament (ALL) reconstruction, with both options aiming to reduce the re-rupture rate relative to traditional quadrupled hamstring grafts.

Objective: To compare, through a prospective and randomized clinical trial, intra and extra-articular ACL reconstruction with ALL using hamstring autograft versus isolated anatomical ACL reconstruction using quintuple or sextuple hamstring autograft.

Methods: 146 patients will be randomized into two groups of 73 patients. Patients included in the study will be evaluated preoperatively and after surgery at 3, 6, 9, 12, and 24 months postoperatively. The primary outcomes will be clinical failure rate and graft rerupture rate. Secondary outcomes will include functional capacity assessed through IKDC, Lysholm KOOS, and Tegner scores, pain using the VAS, as well as stability assessed by digital rolimeter and objective IKDC. Kinesiophobia and anxiety will be measured using the Tampa scale and Anxiety and Depression scale.

Keywords: Rupture, Anterior Cruciate Ligament, Anterior Cruciate Ligament Reconstruction

DETAILED DESCRIPTION:
1. Introduction Arthroscopic reconstruction of the anterior cruciate ligament (ACL) is a well-established procedure known for its superiority over non-surgical treatment of this injury. However, failure rates following ACL reconstruction can vary from 3-6% in some patient cohorts up to 40% in patients at increased risk of re-injury Hamstring autograft are the most commonly used for ACL reconstruction. Considering that the final graft diameter inferior to 8mm is associated to increased failure rate, and that increased intra-articular diameter is considered a protective factor, the preparation of hamstring autografts influences the final outcome. Historically used quadrupled hamstring grafts have been progressively replaced in recent years by quintupled or sextupled graft configurations in order to increase final graft diameter.

   However, instead of using configurations that prioritize increasing the final diameter of hamstring autografts, ACL reconstruction associated with extra-articular reconstruction of the anterolateral ligament (ALL) may be performed using a portion of the gracilis, prioritizing the reconstruction of the ALL rather than increasing the intra-articular graft diameter. The association of the ALL serves two main functions: to decrease rotational instability, which can reach up to 40% in high-risk patients, and to mechanically protect the graft.

   In a comparative analysis pairing patients with similar characteristics, ACL + ALL reconstruction showed significantly lower rerupture rate compared to isolated ACL reconstruction: 3.5% versus 17.4%. In another comparative analysis also pairing patients for similarity, isolated ACL reconstruction with bone-patellar tendon-bone (BTB) autograft showed a 3x higher risk of rerupture compared to ACL + ALL reconstruction with hamstring autografts.

   Thus, the investigators hypothesize that extra-articular reinforcement with ALL reconstruction associated with anatomical ACL reconstruction with hamstring autograft may improve knee stability and help reduce the re-injury rate compared to isolated anatomical reconstruction with quintuple or sextuple hamstrings that prioritize graft diameter, following a well-defined criterion of indication for patients at increased risk of re-injury. In this way, the investigators intend to compare two methods through a randomized clinical trial: intra- and extra-articular reconstruction of the ACL with ALL with hamstring autograft versus isolated anatomical reconstruction of the ACL with quintuple or sextuple hamstring autograft.
2. Hypothesis Anatomical ACL reconstruction associated with extra-articular ALL reconstruction with hamstring autograft will present better functional results, better stability, lower clinical failure rate, and lower graft rupture rate when compared to isolated intra-articular anatomical ACL reconstruction with quintuple or sextuple hamstring autograft.
3. Objectives To compare the functional results, stability, clinical failure rate, and graft rupture rate of individuals undergoing anatomical ACL reconstruction associated with extra-articular ALL reconstruction with hamstring autograft compared to isolated intra-articular anatomical ACL reconstruction with quintuple or sextuple hamstring autograft.
4. Group Formation and Intervention Description

   After randomization, two groups will be formed:

   Group A: Anatomic ACL Reconstruction combined with Extra-Articular Reconstruction with Anterolateral Ligament. The single gracilis strand ALL graft will be passed deep to the iliotibial tract (and superficial to the lateral collateral ligament), entering the tibial tunnel from proximal to distal with its Ethibond terminal portion tied to the tibial terminal portion of the ACL Ethibond with the knee in extension and neutral rotation - without added fixation devices. Wound closure in a layered fashion concludes the procedure.

   Group B: Isolated Intra-Articular Anatomic ACL Reconstruction
5. Patient Evaluation Patients included in the study will be evaluated preoperatively and postoperatively at 3, 6, 9, 12, and 24 months.
6. Return to Sport Criteria All patients will be advised to return to sport only after meeting the following criteria: full range of motion, absence of moderate or severe pain, absence of clinical failure criteria, a minimum of 9 months post-operative period, and completion of FIFA 11+ training for prevention for at least 3 months.
7. Strategies to Improve Adherence and Monitoring Utilization of the Maia Health Tech platform (São Paulo, SP, Brazil), a mobile data collection system with cloud storage and LGPD protection with data anonymization, also using WhatsApp for messaging. Pre-scheduled messages according to the evaluation timeline will assist in patient adherence and monitoring.
8. Circumstances Allowing the Termination of Blinding with Group Revelation Since blinding will occur only for the statistician and partially for data recorders, it will exceptionally be necessary to terminate the blinding.
9. Data Collection Part of the data will be collected in person by people who will have access to knowledge of which group each patient is in. Data will be recorded on the RedCap platform (Vanderbilt, Tennessee).

   Part of the data will be collected remotely, with blinding, using the Maia Health Tech Platform (São Paulo, SP, Brazil), a mobile data collection system with cloud storage and HIPAA-compliant protection with data anonymization, also using WhatsApp for messaging, which will send the following questionnaires to patients: IKDC, Lysholm, KOOS, Tegner, and VAS. One of the investigators will send the patients' phone numbers to the platform so that it can send the data to be collected via WhatsApp through the patient's number. This data will be sent by the Maia Health Tech platform to the RedCap platform autonomously and pre-programmed, without anyone involved in the study intermediating.

   To reduce patient loss during follow-up, the current phone number of the patient, and the phone numbers of two additional close contacts will be collected in case the patient changes their number. The patient will also be instructed to inform the investigator responsible for registering the phone numbers of patients, as well as the Maia Health Tech platform, of any number changes.

   The collected data will be submitted to the RedCap platform. Only the investigators Marcos Vinicius Credidio, Enzo Salviato Mameri, and Thiago Bueno Sanchez will have access to this platform.

   On the RedCap platform, the name, ID, and date of birth of each patient will be included to avoid duplication of records.
10. Statistics A priori Power Analysis - Sample Calculation For the sample size calculation, the G*Power 3.1.9.7 program (http://www.gpower.hhu.de/) was used.

    To compare if there is a difference in the frequencies of variables related to ACL graft rupture rate and clinical failure rate (dichotomous categorical variables) between the two groups of interest, the Chi-Square test was used. For this contingency table, the statistical power calculation considered the following criteria: significance level α of 5%, effect size of 25%, and degree of freedom (df) equal to 1. In a contingency table, the df is calculated as follows: (number of rows - 1) x (number of columns - 1). Considering that the study has two groups and that the variables related to the ACL graft rupture rate and clinical failure rate are dichotomous categorical variables, the calculated degree of freedom was 1. Thus, the sample size calculated for these analyses was 126 individuals. Anticipating a 15% loss of patients during follow-up, 145 patients will be needed to evaluate the graft rupture rate and clinical failure rate as primary outcomes.

    To compare if there is a functional difference through the scores obtained from the IKDC, Lysholm, and KOOS questionnaires (numerical variables) between the two study groups using the t-Student test (parametric) or Mann-Whitney test (non-parametric), using a significance level α of 5%, type β error probability of 20%, an observed power of 80% (1-β), and an effect size of 25%, the total calculated sample size was 506 patients. Anticipating a 15% loss of patients during follow-up, 581 patients will be needed to evaluate functional differences, initially considered secondary outcomes.
11. Statistical Analysis The analysis of quantitative variables will be performed with the calculation of mean, standard deviation, and 95% confidence interval for each estimated point. Secondary variables (categories) will be analyzed through absolute and relative frequency with a 95% confidence interval calculation. Data will be presented in bar graphs and tables for sample characteristics.
12. Interim Analysis and Guidelines for Study Termination A partial analysis will be performed halfway through recruitment with a minimum follow-up of 12 months, and the study will be interrupted if a 30% difference in the primary outcome is observed. The partial analysis will be conducted by a statistician not directly involved in the study, and the decision to terminate the study based on the above criteria will be made by the lead researcher.
13. General, Local Risks, and Adverse Effects The main risks, regardless of the surgical technique used, are as follows: anesthetic risk (e.g., inadvertent punctures, bleeding in venous or spinal anesthesia access, post-spinal anesthesia headache, urinary retention), surgical site infection, swelling and bruising in the knee joint, deep vein thrombosis, pulmonary embolism, neurovascular injuries, unsatisfactory results, and even death (a very rare occurrence but possible in any surgical or anesthetic procedure). The postoperative period presents situations of discomfort inherent to the recovery and rehabilitation of the research participant.

    Adverse effects will be considered any undesirable medical events that the study participant experiences. Range of motion will be evaluated with a goniometer to analyze its loss, and any other signs of clinical problems such as persistent effusion, surgical wound complications, and thrombosis will be documented.

    Serious adverse effects will be considered: unexpected surgical or medication effects resulting in death, life-threatening conditions, requiring hospitalization, resulting in permanent disability, or necessitating surgical intervention for resolution.
14. Benefits for the Patient The benefits to the participant, regardless of the surgical technique used, which are well-established in the literature and routinely performed by the interventionists, include the potential for improved function and reduced pain in the affected limb. Additionally, patients will undergo physical therapy rehabilitation and receive the necessary analgesic support for comfort and well-being. There will be no financial benefit for the patient.
15. Study Justification The study aims to elucidate the best method for preparing hamstring autograft grafts for ACL reconstruction using the same amount of implants in both studied techniques. As these tendons are the most commonly used grafts for ACL reconstruction worldwide, the study's results are expected to have a significant impact on the scientific community, aiding in the better treatment choice for patients.
16. Funding The study will be self-funded.

ELIGIBILITY:
Inclusion Criteria

Patients from the hospital's demand (emergency care and outpatient care) and from CROSS (Center for Regulation of Health Service Offers) who present one or more risk factors will be included:

* Age (Female 14 years - 25 years and Male 16 years - 25 years);
* Pivot-shift test > 2;
* Chronic ACL injury (>12 months);
* Athlete (Tegner Scale ≥ 7);
* Tibial slope > 12 degrees;
* Recurvatum > 5 degrees and < 15 degrees (asymmetric);
* Ligamentous Hypermobility (Beighton Scale > 5).

Non-Inclusion Criteria

* Individuals over 40 years of age will not be included;
* ACL revision;
* PCL injury (grade 2 and 3);
* MCL injury (grade 2 and 3) or (grade 1 with valgus aligned axis);
* CPL injury (grade 2 and 3 according to Fanelli classification);
* Recurrent patellar dislocation;
* Severe chondral lesion (ICRS grade 3 and 4) larger than 1cm2;
* Previous ipsilateral knee surgery;
* Kellgren Lawrence grade 3 or more;
* Autoimmune/rheumatologic inflammatory disease;
* Contralateral knee ligament injury;
* Malalignment > 5 degrees clinical asymmetry between limbs or symmetric > 10 degrees axis deviation to varus (corresponding to > 4 degrees varus between the anatomical axis of the femur and the anatomical axis of the tibia in the clinical examination) or > 10 degrees axis deviation to valgus (corresponding to > 16 degrees valgus between the anatomical axis of the femur and the anatomical axis of the tibia in the clinical examination);
* Graft diameter < 7 mm;
* BMI > 35 or < 18;
* Active or undergoing treatment for malignant neoplasia;
* Pregnancy or suspected pregnancy;
* Psychiatric disorders.

Exclusion Criteria

Leave of absence from work due to disability or reduced income assistance (worker's compensation) whenever one of the investigators considers that the participant may be simulating a worse health condition than reality in order to receive financial assistance with work leave.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical failure rate | Minimum 2 years
  Persistence of pivot shift (grade 1 or higher) in more than one postoperative evaluation compared to the contralateral knee, or a grade 2 or higher pivot shift at any postoperative evaluation.
Graft rupture rate | Minimum 2 years
  Graft rupture will be defined as a graft tear confirmed by magnetic resonance imaging (MRI) or arthroscopy in the presence of any clinical failure criteria.

SECONDARY OUTCOMES:
Functional capacity 1 | Minimum 2 years
  Measured through the Subjective Knee Evaluation Form (IKDC) questionnaire
Functional capacity 2 | Minimum 2 years
  Measured through the Lysholm questionnaire
Functional capacity 3 | Minimum 2 years
  Measured through the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Functional capacity 4 | Minimum 2 years
  Measured through the Tegner questionnaire
Stability 1 | Minimum 2 years
  Measured using a digital rolimeter. Grafts will be classified as functional (side-to-side difference up to 3mm), partially functional (side-to-side difference between 3 and 6mm), and non-functional (side-to-side difference of 6mm or more)
Stability 2 | Minimum 2 years
  Measured using Objective Knee Evaluation Form (IKDC) - Lachman test (grade of 0, 1, 2 and 3)
Stability 3 | Minimum 2 years
  Measured using Objective Knee Evaluation Form (IKDC) - Pivot shift test (grade of 0, 1, 2 and 3)
Stability 4 | Minimum 2 years
  Measured Objective Knee Evaluation Form (IKDC) - Anterior drawer test (grade of 0, 1, 2 and 3)
Kinesiophobia | Minimum 2 years
  Measured using the Tampa Scale
Anxiety Scale | Minimum 2 years
  Measured using the Anxiety and Depression Scale
Pain Scale | Minimum 2 years
  Measured using the Visual Analog Scale (VAS) - (score from 0 to 10 )

CONTACTS AND LOCATIONS:
Overall Officials: MARCOS VINICIUS CREDIDIO, Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Sao Paulo Hospital, São Paulo, São Paulo
  - Parelheiros Hospital, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
Protocolo de Estudo